CLINICAL TRIAL: NCT04379245
Title: Study of the Attack Rate of COVID-19 Infection in Patients Infected With HIV and/or on Pre-exposure Prophylaxis (PrEP) and Possible Impact of Treatment With an HIV Protease Inhibitor
Brief Title: COVID-19 Infection in Patients Infected With HIV and/or on PrEP
Acronym: COVIDHIVPrEP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2020_002
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: HIV; Pre-exposure Prophylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data research, database analysis — Extraction of virological data at the virology laboratory (date, SARS-COV2 PCR result, identification number, sex, date of birth) (Excel file)
  * Extraction of demographic and viro-immunological data from patients infected with HIV and on PrEP followed at the Hospices Civils de Lyon, France, over the period concerned (Access extraction)
  * Data crossing (Excel / Access) and statistical analysis
  * Calculation of the positivity rate per calendar period (= number of diagnosed cases / number of patients tested) and the attack rate per calendar period (number of diagnosed cases / number of people exposed (= active file of patients followed reduced by the number already known to be positive)).

SUMMARY:
The SARS-CoV-2 epidemic was declared as a global pandemic by the WHO on March 12, 2020. France is affected with approximately 120,000 biologically confirmed cases, as of April 30, 2020, a figure probably very underestimated. Its distribution in different populations, in particular immunocompromised, has not yet been measured. The in vitro efficacy of lopinavir coupled with ritonavir, an HIV protease inhibitor, on SARS-CoV, responsible for SARS has been discussed and this therapeutic combination is currently being evaluated in patients infected with COVID-19. The possible protective role of treatment with Lopinavir / ritonavir or another HIV protease inhibitor has not been studied.

In addition, patients receiving HIV pre-exposure prophylaxis (PrEP) share certain epidemiological and behavioral characteristics with HIV-infected patients.

The objective was to carry out an epidemiological study aimed at determining the attack rate of COVID-19 infection in patients infected with HIV and or on PrEP and to analyze this attack rate according to the characteristics of these 2 populations and in particular the existence or not of an antiretroviral treatment comprising Lopinavir / Ritonavir or another inhibitor of the HIV protease.

Cross-referencing of Virology Laboratory data (positive or negative screening) and clinical-biological data can be easily carried out using a unique identification number in the 2 software programs and will allow an almost exhaustive epidemiological analysis in 2 well identified populations.

ELIGIBILITY:
Inclusion Criteria:

* HIV patients in Hospices Civils de Lyon
* on-PrEP patients in Hospices Civils de Lyon

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two populations will be studied:
  * HIV patients in Hospices Civils de Lyon
  * on PrEP patients in Hospices Civils de Lyon
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Covid attack rate | During hospitalisation for Covid symptoms: one week (max 2 weeks) after symptoms initiation
  Cross-referencing of Virology Laboratory data (positive or negative screening) and clinical-biological data using the unique identification number in the 2 databases. This cross-checking of files will allow an almost exhaustive epidemiological analysis in 2 well identified populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No